CLINICAL TRIAL: NCT02449278
Title: The Palliative Benefit of Involved-site Radiotherapy Following Effective Chemotherapy for Patients With Advanced-stage Diffuse Large B-cell Lymphoma: Wuhan University Cancer Center - NHL04 Trial
Brief Title: The Palliative Benefit of Involved-site Radiotherapy for Patients With Advanced-stage Diffuse Large B-cell Lymphoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wuhan University (Other)
Responsible Party: Principal Investigator, Di Deng, Director,Clinical Research, Wuhan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WUCC-NHL04 Trial
Record Dates: First submitted 2015-05-07; First posted 2015-05-20 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-12

CONDITIONS: Diffuse Large B-cell Lymphoma
Keywords: advanced-stage DLBCL; ISRT; chemotherapy
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Cyclophosphamide; Doxorubicin; Vincristine; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ISRT group (Experimental): Six cycles Chemotherapy (cyclophosphamide 750mg/square meter on day 1 + doxorubicin 50mg/square meter on day 1 + vincristine 1.4mg/square meter on day 1 (up to a maximal dose of 2 mg) + prednisone 60mg/square meter on day 1 through 5, repeated at 21-day intervals) .
  Consolidation involved-site radiotherapy (ISRT) following in patient with complete or partial response beginning 1 month after last cycle of chemotherapy.
  Interventions: Radiation: Consolidation involved-site radiotherapy (ISRT); Drug: cyclophosphamide; Drug: doxorubicin; Drug: vincristine; Drug: prednisone
- IFRT group (Active Comparator): Six cycles Chemotherapy (cyclophosphamide 750mg/square meter on day 1 + doxorubicin 50mg/square meter on day 1 + vincristine 1.4mg/square meter on day 1 (up to a maximal dose of 2 mg) + prednisone 60mg/square meter on day 1 through 5, repeated at 21-day intervals).
  Consolidation involved-field radiotherapy (IFRT) following in patient with complete or partial response beginning 1 month after last cycle of chemotherapy.
  Interventions: Radiation: Consolidation involved-field radiotherapy (IFRT); Drug: cyclophosphamide; Drug: doxorubicin; Drug: vincristine; Drug: prednisone

INTERVENTIONS:
Radiation: Consolidation involved-site radiotherapy (ISRT) — 6 cycles modern CHOP chemotherapy followed consolidation involved-site radiotherapy (ISRT).
  Involved-site radiotherapy (ISRT) is based on defining the site of gross disease before chemotherapy, the GTV and using a CT-based volume with an expansion to form a CTV in the cranio-caudal direction.
  The general dose had been guided that 30-36Gy in 15~18 fractions of 2 Gy 5 days per week was managed for patients with complete response (CR) after chemotherapy and 40-50Gy in 20~25 fractions of 2 Gy 5 days per week for partial response (PR).
  Arms: ISRT group
Radiation: Consolidation involved-field radiotherapy (IFRT) — 6 cycles modern CHOP chemotherapy followed consolidation involved-field radiotherapy (IFRT).
  Radiotherapy field of IFRT defined by CALGB is encompassed the prechemotherapy gross tumor.
  The general dose had been guided that 30-36Gy in 15~18 fractions of 2 Gy 5 days per week was managed for patients with complete response (CR) after chemotherapy and 40-50Gy in 20~25 fractions of 2 Gy 5 days per week for partial response (PR).
  Arms: IFRT group
Drug: cyclophosphamide — Patients in both arms will be given cyclophosphamide chemotherapy
Drug: doxorubicin — Patients in both arms will be given doxorubicin chemotherapy
Drug: vincristine — Patients in both arms will be given vincristine chemotherapy
Drug: prednisone — Patients in both arms will be given prednisone chemotherapy

SUMMARY:
The standard treatment approach for patients with stage III-IV DLBCL is combination chemotherapy. Receipt of consolidation radiotherapy (RT) after effective chemotherapy was associated with improved in-field control and event-free survival. However, it is uncertain for the radiotherapy field size to treat for these patients after chemotherapy. Involved-field radiotherapy (IFRT) after effective chemotherapy is a common strategy for patients with stage III-IV DLBCL. There is not a clinical trial to research whether the sequential narrowed radiotherapy field size (involved-site radiotherapy, ISRT) can obtain the same efficacy as IFRT and decrease toxicities related to radiotherapy.

DETAILED DESCRIPTION:
Diffuse large B-cell lymphoma (DLBCL) is the most common subtype of non-Hodgkin lymphoma. Approximately 50% of patients present with stage III-IV disease at diagnosis. The standard treatment approach for these patients is combination chemotherapy. the role of radiation therapy (RT) after effective system therapy in stage III-IV DLBCL (advanced-stage DLBCL) is controversial. The recommended approaches for patients with stage III-IV disease by The National Comprehensive Cancer Network (NCCN) are that consolidation RT is managed for patients who achieved a complete response (CR) to chemotherapy and palliative RT for patients with partial response (PR) after chemotherapy. However, it is uncertain for the radiotherapy field size to treat for these patients after chemotherapy.

Some benefits of consolidation RT after chemotherapy exist for patients with advanced-stage DLBCL. One of the important aims of treatment for these patients is the improvement of event-free survival (EFS). After patients receive chemotherapy alone, the most common site of disease recurrence is at sites of initial disease involvement. The complications related to chemotherapy, including second malignancies and other non-neoplastic late events, were needed to emphasize for those patients managed with more cycles' regimens alone to increase the efficacy of patients with advanced-stage DLBCL. Receipt of consolidation RT was associated with improved in-field control and EFS though no difference in overall survival (OS) when compared to patients without consolidation RT. Several randomized and retrospective studies demonstrated that the EFS (even the OS) can be improved by consolidation RT for patients with advanced-stage DLBCL after CHOP or CHOP-like chemotherapy. The patients randomized among those diagnosed initially with bulky disease (>10 cm), those achieving CR or PR after chemotherapy, and even those in stage IV with bone marrow involved.

The complications related to consolidation RT also need to be additionally explored for those patients since the efficacy of advanced-stage DLBCL has improved by combined-modality therapy (CMT). Especially, considerable difficulties in the continuous salvage options are unavoidable because of the risk of blood cell production disorders associated to extensive-field radiotherapy. Consolidation involved-field radiotherapy (IFRT) after effective chemotherapy is common palliative strategy for patients with advanced-stage DLBCL. The morbidity of treatment may be decreased further by RT with the radiation field size reduction. Involved-site radiotherapy (ISRT), based on a modified involved field, aims to reduce the radiation volume treated and the probability of late effects. Its radiation targets include a gross tumor volume (GTV), a clinical target volume (CTV), and a planning target volume (PTV), which were defined in International Commission on Radiation Units and Measurements Report (ICRU) 50. This is based on defining the site of gross disease before chemotherapy, the GTV and using a CT-based volume with an expansion to form a CTV in the cranio-caudal direction. There is not a clinical trial to research whether the sequential narrowed radiotherapy field size (involved-site radiotherapy, ISRT) can obtain the same efficacy as IFRT and decrease toxicities related to radiotherapy.

To evaluate the differences between IFRT and ISRT in the efficacy and complications related to consolidation RT for patients with advanced-stage DLBCL who achieved effective chemotherapy. The CTV of ISRT is defined as the region including the prechemotherapy volume of disease with 1.5 cm margin expanded cranio-caudally in the direction of potential lymphatic spread. The CTV should not extend into air in the transverse plane and should be limited in the involved lymph node region defined by the Cancer and Leukemia Group B (CALGB). The PTV is then extended from CTV by adding the necessary margin for setup error and organ motion.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female aged range from 18 years to 65 years.
* Eastern Cooperative Oncology Group(ECOG) performance status of 0 or 1.
* All patients had histologically confirmed Diffuse large B-cell lymphoma.
* Advanced-stage DLBCL patients at newly diagnosed or recurrent without RT in initial management.
* Adequate organ function.
* Negative pregnancy test.
* Signed informed consent document on file.

Exclusion Criteria:

* Woman who were pregnant or lactating.
* With severe local infection or general infective disease.
* Primary lymphoma in special organ including cuticula, center never system, gastrointestinal tract, testicle, and lung.
* With other second primary malignancy except cutaneum carcinoma.
* Being or planning to participate in other study.
* Any patient who in the opinion of the investigator should not participate in the study.

Withdrawal Criteria:

* Patient are free to withdrawal completely from the study at any time upon request.
* Patient in the study may be stopped with the patient agreement at any time at the discretion of investigator.
* In-field progression on irradiation ongoing.
* Poor tolerability adverse events in the period of chemotherapy or irradiation after enrolled in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-10; Primary Completion 2019-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival - PFS | from the date of diagnosis to the date of treatment failure or death from any cause, whichever occurs first, Assessed up to 100 months.
  Treatment failure was defined as any recurrence of non-Hodgkin lymphoma.
Adverse events with grade 3 or 4 - AEs | The time from the day of treatment to the day of the first documented disease progression or death from any cause, Assessed up to 24 months.
  Toxicity was scored according to the toxicity scale of the National Cancer Institute Common Terminology Criteria for Adverse Events 3.0.

SECONDARY OUTCOMES:
Overall survival - OS | From the initial diagnosis of follicular lymphoma to death from any cause, Assessed up to 120 months.
Rate of in-field progression | From the start of RT to the first documented disease progression within the radiotherapy field, Assessed up to 60 months.
Rate of out-field progression | From the start of RT to the first documented disease progression outside the radiotherapy field, Assessed up to 60 months.
Rate of regional failure | From the start of RT to the first documented disease progression outside of ISRT field but within the involved region defined as CALGB, Assessed up to 60 months.

CONTACTS AND LOCATIONS:
Locations (1):
- DiDeng, Wuhan, Hubei, China